CLINICAL TRIAL: NCT01018784
Title: A Phase 1 Study of MORAb-009 in Patients With Solid Tumor
Brief Title: A Study of MORAb-009 in Patients With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAB-009-J081-102
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Cancer; Mesothelin-positive
Keywords: Cancer; Mesothelin-positive
MeSH Terms: conditions — Neoplasms | interventions — amatuximab

ARMS (1):
- MORAb-009 (Experimental)
  Interventions: Drug: MORAb-009

INTERVENTIONS:
Drug: MORAb-009 — MORAb-009 is intravenously administered to patients with solid tumor once a week for 4 weeks as 1 cycle.

SUMMARY:
MORAb-009 is intravenously administered to patients with solid tumor once a week for 4 weeks as 1 cycle in order to investigate dose-limiting toxicity and estimate maximum tolerated dose.

ELIGIBILITY:
Inclusion criteria;

1. Japanese male and female patients aged from 20 to less than 80 years at obtaining informed consent
2. Patient with histologically or cytologically diagnosed solid tumor
3. Patient who is mesothelin-positive confirmed by immunohistochemistry (IHC) (except for pancreatic cancer and mesothelioma that mesothelin-positive is frequently reported)
4. Patient with solid tumor who is non responder to or resistant to standard therapy and has no other appropriate treatment
5. Performance Status (PS) is 0 to 1 by Eastern Cooperative Oncology Group ECOG criteria

Exclusion criteria

1. Brain metastasis presenting clinical symptoms or requiring medical treatment
2. Serious and systemic infection requiring medical treatment
3. History of hypersensitivity to protein formulations including monoclonal antibody
4. With active multiple carcinoma (except for carcinoma in situ and intramucosal carcinoma)
5. With celomic fluid (pleural effusion or ascites) uncontrolled by drainage, or with a large volume of celomic fluid

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To investigate dose-limiting toxicity and estimate maximum tolerated dose. | 4 Weeks

SECONDARY OUTCOMES:
The best overall response rate in the RECIST evaluation and the preliminary evaluation calculating the frequency of Completed response and Partial Response. | During Study

CONTACTS AND LOCATIONS:
Overall Officials: Chifumi Kitamura, Study Director — Morphotek Clinical Development Section, JAC PCU
Locations (1):
- Sayama-shi, Osaka, Japan

REFERENCES:
- [Derived] Fujisaka Y, Kurata T, Tanaka K, Kudo T, Okamoto K, Tsurutani J, Kaneda H, Okamoto I, Namiki M, Kitamura C, Nakagawa K. Phase I study of amatuximab, a novel monoclonal antibody to mesothelin, in Japanese patients with advanced solid tumors. Invest New Drugs. 2015 Apr;33(2):380-8. doi: 10.1007/s10637-014-0196-0. Epub 2014 Dec 12. PMID 25502863